CLINICAL TRIAL: NCT06030999
Title: Three Arms, Randomized, Double-blind Controlled Trial Of Prevention And Treatment On Obesity And Weight Management By Oral Supplementation Of Probiotics And Prebiotics
Brief Title: The Prevention And Treatment On Obesity And Weight Management By Oral Supplementation Of Probiotics And Prebiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Precision Health Food Technology Co. Ltd., (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 23-SM-08-WL-001
Record Dates: First submitted 2023-09-03; First posted 2023-09-11 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Overweight and Obesity
Keywords: Probiotics; Prebiotics; Wonderlab
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study product A (Wonderlab wonder4shape) (Active Comparator): 2g/bottle, containing the following probiotics total dosage 2.0*1010 CFU:
  * CECT7527, CECT7528, CECT7529
  * Maltodextrin
  * Lactobacillus acidophilus
  * Fructose oligosaccharides
  * Grapefruit, Lemon and Apple powder
  Interventions: Dietary Supplement: Study product A (Wonderlab wonder4shape)
- Study product B (Wonderlab wonder4shape) (Active Comparator): 2g/bottle, containing the following probiotics total dosage 1.0*1010 CFU:
  * Maltodextrin
  * Lactobacillus acidophilus
  Interventions: Dietary Supplement: Study product B (Wonderlab wonder4shape)
- Study product C (placebo) (Placebo Comparator): 2g/bottle, containing the following ingredients:
  * Maltodextrin
  * Grapefruit powder
  * Lemon powder
  Interventions: Dietary Supplement: Study product C (placebo)

INTERVENTIONS:
Dietary Supplement: Study product A (Wonderlab wonder4shape) — Participants in this arm need to consume one bottle (2g) of this product once a day for 10 weeks
  Arms: Study product A (Wonderlab wonder4shape)
Dietary Supplement: Study product B (Wonderlab wonder4shape) — Participants in this arm need to consume one bottle (2g) of this product once a day for 10 weeks
  Arms: Study product B (Wonderlab wonder4shape)
Dietary Supplement: Study product C (placebo) — Participants in this arm need to consume one bottle (2g) of this product once a day for 10 weeks
  Arms: Study product C (placebo)

SUMMARY:
The goal of this interventional study is to test whether consumption of Wonderlab probiotics with prebiotics could improve obesity and overweight in Chinese people who are aged 25-45 and overweight. The main question it aims to answer is:

- whether the weight of participants can be lost after 10 weeks' intervention

150 participants will be randomized into 3 study groups (50 each group) in the two study sites, who will consume assigned product according to instructions for 10 weeks. Three site visits will be made for each participant and all relevant clinical data will be captured and recorded into CTMS(Clinical Trial Management System) for statistical analysis.

Researchers will compare the three groups to conclude whether the Wonderlab study product can improve obesity and overweight over placebo product.

ELIGIBILITY:
Inclusion Criteria:

* Chinese males or females, age between 25-45;
* Overweight population: BMI 24-27.9 & obesity population: BMI >=28;
* Blood lipids in high potential risks but without medication:TG > 5mmol/L or LDL >= 3.4 mmol/L or TC >= 5.2 mmol/L.
* Understand the test procedure, read, and sign an appropriate Informed Consent Form indicating their willingness to participate;
* Agree to avoid medication treatment for weight management, including blood lipids and sugar control.

Exclusion Criteria:

* Have used any medication for weight management at least one month before this study.
* Subject having done plastic surgery for weight management.
* Be involved in any aspect of test administration, i.e., evaluating or overseeing activities related to product.
* Have participated in any clinical study involving the test sites within the previous 6 months, or is subject participating in any clinical study concurrently.
* Have a history of any type of metabolic syndrome, including but not limited to any type of diabetes, obesity and heart disease.
* Have a history of any disease or the presence of health condition on the study sites that the Investigator feels would interfere with the study.
* Be taking antihistamines (> 3x/week) or anti-inflammatory (> 8x/week) on a regular basis, or has the subject taken systemic or topical steroidal medications within 4 weeks of study enrolment.
* Have any of the following conditions or factors that the investigator believes may affect the response of the skin or the interpretation of the test results, including, but not limited to, pregnancy, lactation and hepatitis.
* Have any cuts/abrasions on the test site at baseline.
* The subject is an employee of sponsor or the site conducting the study.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2023-12-02 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Change of Weight | baseline day 0, day 70
  Change of Weight in Kg by Inbody S10 from baseline to 10 weeks

SECONDARY OUTCOMES:
Blood lipids - Total Cholesterol Level | baseline day 0, day 35, day 70
  Blood lipids - Total Cholesterol level of blood test in mmol/L and range of 0.56-17mmol/L for each visit interval
Blood Sugar Level | baseline day 0, day 35, day 70
  Blood sugar level of blood test in mmol/L and range of 3.9-6.1mmol/L
Blood hormone - Leptin level | baseline day 0, day 35, day 70
  Blood hormone - Leptin level of blood test in ng/mL and range 0.5-15.2ng/mL
Blood hormone - Adiponectin level | baseline day 0, day 35, day 70
  Blood hormone - Adiponectin level of blood test in ug/mL and range of 2-37ug/mL
Blood inflammation | baseline day 0, day 35, day 70
  Blood inflammation (Zonulin, ApoB-48, hsCRP, LPS, sCD14, IL-6, MCP-1, Angptl4)

CONTACTS AND LOCATIONS:
Overall Officials: Hongwei Guo, MD, Principal Investigator — Shanghai Fudan University, School of Public Health; Weixing Wang, MD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (2):
- China (2):
  - SPRIM Central Lab, Shanghai, Shanghai Municipality
  - Ligang Hospital, Jinhua, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aoun A, Darwish F, Hamod N. The Influence of the Gut Microbiome on Obesity in Adults and the Role of Probiotics, Prebiotics, and Synbiotics for Weight Loss. Prev Nutr Food Sci. 2020 Jun 30;25(2):113-123. doi: 10.3746/pnf.2020.25.2.113. PMID 32676461
- [Background] Guirro M, Costa A, Gual-Grau A, Herrero P, Torrell H, Canela N, Arola L. Effects from diet-induced gut microbiota dysbiosis and obesity can be ameliorated by fecal microbiota transplantation: A multiomics approach. PLoS One. 2019 Sep 23;14(9):e0218143. doi: 10.1371/journal.pone.0218143. eCollection 2019. PMID 31545802
- [Background] Gill VJS, Soni S, Shringarpure M, Anusheel, Bhardwaj S, Yadav NK, Patel A, Patel A. Gut Microbiota Interventions for the Management of Obesity: A Literature Review. Cureus. 2022 Sep 19;14(9):e29317. doi: 10.7759/cureus.29317. eCollection 2022 Sep. PMID 36161997
- [Background] Hill C, Guarner F, Reid G, Gibson GR, Merenstein DJ, Pot B, Morelli L, Canani RB, Flint HJ, Salminen S, Calder PC, Sanders ME. Expert consensus document. The International Scientific Association for Probiotics and Prebiotics consensus statement on the scope and appropriate use of the term probiotic. Nat Rev Gastroenterol Hepatol. 2014 Aug;11(8):506-14. doi: 10.1038/nrgastro.2014.66. Epub 2014 Jun 10. PMID 24912386
- [Background] Gibson GR, Hutkins R, Sanders ME, Prescott SL, Reimer RA, Salminen SJ, Scott K, Stanton C, Swanson KS, Cani PD, Verbeke K, Reid G. Expert consensus document: The International Scientific Association for Probiotics and Prebiotics (ISAPP) consensus statement on the definition and scope of prebiotics. Nat Rev Gastroenterol Hepatol. 2017 Aug;14(8):491-502. doi: 10.1038/nrgastro.2017.75. Epub 2017 Jun 14. PMID 28611480
- [Background] Swanson KS, Gibson GR, Hutkins R, Reimer RA, Reid G, Verbeke K, Scott KP, Holscher HD, Azad MB, Delzenne NM, Sanders ME. The International Scientific Association for Probiotics and Prebiotics (ISAPP) consensus statement on the definition and scope of synbiotics. Nat Rev Gastroenterol Hepatol. 2020 Nov;17(11):687-701. doi: 10.1038/s41575-020-0344-2. Epub 2020 Aug 21. PMID 32826966
- [Background] Arora T, Sharma R. Fermentation potential of the gut microbiome: implications for energy homeostasis and weight management. Nutr Rev. 2011 Feb;69(2):99-106. doi: 10.1111/j.1753-4887.2010.00365.x. PMID 21294743
- [Background] Lee HY, Park JH, Seok SH, Baek MW, Kim DJ, Lee KE, Paek KS, Lee Y, Park JH. Human originated bacteria, Lactobacillus rhamnosus PL60, produce conjugated linoleic acid and show anti-obesity effects in diet-induced obese mice. Biochim Biophys Acta. 2006 Jul;1761(7):736-44. doi: 10.1016/j.bbalip.2006.05.007. Epub 2006 May 20. PMID 16807088
- [Background] Martin FP, Wang Y, Sprenger N, Yap IK, Lundstedt T, Lek P, Rezzi S, Ramadan Z, van Bladeren P, Fay LB, Kochhar S, Lindon JC, Holmes E, Nicholson JK. Probiotic modulation of symbiotic gut microbial-host metabolic interactions in a humanized microbiome mouse model. Mol Syst Biol. 2008;4:157. doi: 10.1038/msb4100190. Epub 2008 Jan 15. PMID 18197175
- [Background] Guazzelli Marques C, de Piano Ganen A, Zaccaro de Barros A, Thomatieli Dos Santos RV, Dos Santos Quaresma MVL. Weight loss probiotic supplementation effect in overweight and obesity subjects: A review. Clin Nutr. 2020 Mar;39(3):694-704. doi: 10.1016/j.clnu.2019.03.034. Epub 2019 Apr 3. PMID 30987812
- [Background] Bosch M, Fuentes MC, Audivert S, Bonachera MA, Peiro S, Cune J. Lactobacillus plantarum CECT 7527, 7528 and 7529: probiotic candidates to reduce cholesterol levels. J Sci Food Agric. 2014 Mar 15;94(4):803-9. doi: 10.1002/jsfa.6467. Epub 2013 Dec 4. PMID 24186773
- [Background] Kim GB, Yi SH, Lee BH. Purification and characterization of three different types of bile salt hydrolases from Bifidobacterium strains. J Dairy Sci. 2004 Feb;87(2):258-66. doi: 10.3168/jds.S0022-0302(04)73164-1. PMID 14762068
- [Background] Begley M, Hill C, Gahan CG. Bile salt hydrolase activity in probiotics. Appl Environ Microbiol. 2006 Mar;72(3):1729-38. doi: 10.1128/AEM.72.3.1729-1738.2006. No abstract available. PMID 16517616
- [Background] Verhoog S, Taneri PE, Roa Diaz ZM, Marques-Vidal P, Troup JP, Bally L, Franco OH, Glisic M, Muka T. Dietary Factors and Modulation of Bacteria Strains of Akkermansia muciniphila and Faecalibacterium prausnitzii: A Systematic Review. Nutrients. 2019 Jul 11;11(7):1565. doi: 10.3390/nu11071565. PMID 31336737
- [Background] Hills RD Jr, Pontefract BA, Mishcon HR, Black CA, Sutton SC, Theberge CR. Gut Microbiome: Profound Implications for Diet and Disease. Nutrients. 2019 Jul 16;11(7):1613. doi: 10.3390/nu11071613. PMID 31315227